CLINICAL TRIAL: NCT04917237
Title: Non-disabling Ischemic Cerebrovascular Event With Apathy: A Prospective Registry Trail
Brief Title: Non-disabling Ischemic Cerebrovascular Event With Apathy
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Bingying Du, Professor, Changhai Hospital
Other Study IDs: NICE-A
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Apathy; Minor Stroke; Transient Ischemic Attack; Stroke
Keywords: Apathy; minor stroke; Transient Ischemic Attack; Stroke
MeSH Terms: conditions — Lethargy; Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The burden of non-disabling ischemic cerebrovascular events (NICE) is significantly increased. However, few previous studies have focused on affective impairment after transient ischemic attack (TIA) and minor stroke. Stroke survivors are often described as apathetic. Even though post-stroke apathy (PSA) affects one in three stroke patients,it has not hitherto received much attention. NICE-A is a prospective study aimed to explore the association between baseline apathy and probable incident stroke in a population-based sample of TIA and minor stroke adults.

DETAILED DESCRIPTION:
Transient ischemic attack (TIA) and acute minor ischemic stroke, are common and may leave impermanent or mild neurological deficit, they are termed as non-disabling ischemic cerebrovascular disease (NICE). TIA and minor stroke exhibit the common substantial risk factors for early stroke recurrence and epidemiological characteristic, with approximately 10 to 20% of patients having a stroke within 3 months after the index event.

Previous studies has shown that post-stroke apathy (PSA) affects one in three stroke patients, which is consistently associated with a worse level of functional recovery, poorer overall health and poorer quality of life. However, still little is known about the development of TIA and minor stroke patients with apathy. Thus, it is imperative to find the relationships between baseline PSA and probable incident stroke in these patients.

NICE is an attractive researching area globally. According to the large quantities of NICE patients in China and the low standardized therapeutic rate, the awareness of TIA and minor stroke is largely insufficient. The purpose of the present NICE-A study is to establish the prevalence, predictors and evolution of symptoms of PSA in TIA and minor stroke patients during the first post-stroke year.

ELIGIBILITY:
Inclusion Criteria:

≥18 years old Onset of a minor stroke (National Institute of Health stroke scale, NIHSS≤3) and TIA elapsed time from last episode to registry <1 month

Exclusion Criteria:

patients who refused to participate in the research, and patients who failed to complete the follow-up protocol.

patients with malignant tumors, or patients with severe liver or kidney disease, whose life expectancy is less than 1 year.

patients who received endovascular or thrombolytic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults patients (≥18 years) within 1 month of onset of a minor stroke (National Institute of Health stroke scale, NIHSS≤3) and TIA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Death | 1 month
  Death from any cause
Death | 3 months
  Death from any cause
Death | 6 months
  Death from any cause
Death | 12 months
  Death from any cause
Stroke recurrence | 1 month
  Ischemic stroke
Stroke recurrence | 3 months
  Ischemic stroke
Stroke recurrence | 6 months
  Ischemic stroke
Stroke recurrence | 12 months
  Ischemic stroke

SECONDARY OUTCOMES:
Hemorrhagic stroke | 1 month
  Cerebral hemorrhage and subaraclmoid hemorrhage
Hemorrhagic stroke | 3 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Hemorrhagic stroke | 6 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Hemorrhagic stroke | 12 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Functional outcome | 1 month
  Modified Rankin Scale ≥3
Functional outcome | 3 months
  Modified Rankin Scale ≥3
Functional outcome | 6 months
  Modified Rankin Scale ≥3
Functional outcome | 12 months
  Modified Rankin Scale ≥3

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Bi, MD, PhD, Principal Investigator — Department of Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided